CLINICAL TRIAL: NCT02743286
Title: Sedentary Behavior Interrupted - A Pilot Study of Acute Interventions on Prolonged Sitting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Dorothy Sears, Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 150509
Record Dates: First submitted 2016-03-30; First posted 2016-04-19 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Sedentary Lifestyle
Keywords: sedentary behavior; sitting; feasibility; endothelial function; metabolism
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control condition (Protocol A) (No Intervention): Following a one-hour sitting run-in period, participants will sit for a 5-hour period including a mid-point bathroom break.
- Frequent sit-to-stands (Protocol B) (Experimental): Following a 1-hour sitting run-in period, participants will sit for a 5-hour period including 15 2-minute standing interruptions, 3 per hour, and a mid-point bathroom break.
  Interventions: Behavioral: Frequent sit-to-stands
- Walking breaks (Protocol C) (Experimental): Following a 1-hour sitting run-in period, participants will sit for a 5-hour period including 5 2-minute walking interruptions, 3 per hour, and a mid-point bathroom break.
  Interventions: Behavioral: Walking breaks
- Stand More (Protocol D) (Experimental): Following a 1-hour sitting run-in period, participants will sit for a 5-hour period including 5 10-minute standing breaks, 1 per hour, and a mid-point bathroom break.
  Interventions: Behavioral: Stand more

INTERVENTIONS:
Behavioral: Frequent sit-to-stands — Participants will visit the clinic for a 6-hour monitoring period. Following a 1-hour sitting run-in period, participants will sit for an additional 5-hour period including 15 2-minute standing interruptions, 3 per hour. Baseline, mid-point, and end-of-visit bathroom breaks for urine sample collection will be conducted, with additional bathroom breaks allowed as needed.
  Other Names: Protocol B
  Arms: Frequent sit-to-stands (Protocol B)
Behavioral: Walking breaks — Participants will visit the clinic for a 6-hour monitoring period. Following a 1-hour sitting run-in period, participants will sit for an additional 5-hour period including 5 2-minute walking interruptions, 3 per hour. Baseline, mid-point, and end-of-visit bathroom breaks for urine sample collection will be conducted, with additional bathroom breaks allowed as needed.
  Other Names: Protocol C
  Arms: Walking breaks (Protocol C)
Behavioral: Stand more — Participants will visit the clinic for a 6-hour monitoring period. Following a 1-hour sitting run-in period, participants will sit for an additional 5-hour period including 5 10-minute standing interruptions, 1 per hour. Baseline, mid-point, and end-of-visit bathroom breaks for urine sample collection will be conducted, with additional bathroom breaks allowed as needed.
  Other Names: Protocol D
  Arms: Stand More (Protocol D)

SUMMARY:
Sedentary behavior, characterized by excess sitting time during waking hours, is detrimental to health and increases cardiometabolic disease risk, independent of moderate-to-vigorous physical activity. The mechanisms that mediate this are unknown and there are no evidence-based methods known for effectively intervening on sedentary behavior. The consequences of prolonged sitting time are of particular interest in older adults as sedentary behavior and cardiometabolic disease risk both increase with aging and moderate-to-vigorous physical activity may not be feasible. This pilot study will assess interventions for sedentary older adults designed to interrupt prolonged sitting time. Interrupting sitting time through sit-to-stand transitions, and standing and walking breaks increases muscle use and blood flow in the lower parts of the body. Thus, the investigators believe that frequent sit-to-stand interruptions of sitting time are the most efficacious sedentary behavior interventions, compared to simply reducing sitting time or less frequent walking breaks, for improving health outcomes and healthy aging. The investigators hypothesize that frequency of sit-to-stands during a 5-hour sitting period will result in health benefits that can be observed with a simple 2-minute standing interruption, and that this will be associated with improvements in metabolism and endothelial function. This pilot, 10-participant study will 1) generate preliminary data for a revised Program Project Grant application to the National Institute of Aging (NIA) that focuses on postmenopausal women, the fastest growing aged population with high life-time risk of cardiometabolic risk. This pilot study will inform sitting interruption modality design for two projects in the investigators' Program Project Grant application: "Project 1: Sedentary Behavior Interrupted: A randomized crossover treatment trial of acute effects on biomarkers of healthy aging in the laboratory (86 participants)" and "Project 2: Sedentary Behavior Interrupted: A randomized trial of 6 month effects on biomarkers of healthy aging and physical functioning in the real world (660 participants)." The current design of this pilot study is enhanced by and responsive to feedback from our initial NIA submission. This pilot study will increase our knowledge about how sedentary behavior and sitting interruption interventions influence healthy aging in postmenopausal women.

DETAILED DESCRIPTION:
Sedentary behavior, characterized by excess sitting time during waking hours, is detrimental to health and increases cardiometabolic disease (e.g., type 2 diabetes) risk, independent of moderate-to-vigorous physical activity. The mechanisms that mediate this are unknown and there are no evidence-based methods known for effectively intervening on sedentary behavior. The consequences of prolonged sitting time are of particular interest in older adults as sedentary behavior and cardiometabolic disease risk both increase with aging and moderate-to-vigorous physical activity may not be feasible. The investigators propose pilot and feasibility testing of interventions for sedentary older adults that are designed to interrupt prolonged sitting time. Interrupting sitting time through sit-to-stand transitions, and standing and walking breaks increases muscle use and blood flow in the lower parts of the body. Thus, the investigators believe that frequent sit-to-stand interruptions of sitting time are the most efficacious sedentary behavior interventions, compared to simply reducing sitting time or less frequent walking breaks, for improving health outcomes and healthy aging. The investigators hypothesize that frequent sit-to-stands during a 5-hour sitting period will result in health benefits that can be observed with a simple 2-minute standing interruption, and that this will be associated with improvements in metabolism and endothelial function. This pilot, 10-participant study will 1) generate preliminary data for a revised Program Project Grant application to the National Institute of Aging (NIA) that focuses on postmenopausal women, the fastest growing aged population with high life-time risk of cardiometabolic risk. This pilot study will inform sitting interruption modality design for two projects in the investigators' Program Project Grant application: "Project 1: Sedentary Behavior Interrupted: A randomized crossover treatment trial of acute effects on biomarkers of healthy aging in the laboratory (86 participants)" and "Project 2: Sedentary Behavior Interrupted: A randomized trial of 6 month effects on biomarkers of healthy aging and physical functioning in the real world (660 participants)." The current design of this pilot study is enhanced by and responsive to feedback from our initial NIA submission. This pilot study will increase our knowledge about how sedentary behavior and sitting interruption interventions influence healthy aging in postmenopausal women.

SPECIFIC AIM The deleterious health consequences of too much sitting are independent of moderate-to-vigorous physical activity. Understanding the health consequences of sitting time is particularly relevant for older adults who are extremely sedentary and at high risk of several chronic diseases that have been linked with sitting time, including type 2 diabetes. Interestingly, sedentary behavior is least studied among older adults who may benefit the most from reducing sitting time. Reducing uninterrupted sitting time in older adults is a research priority because the pervasiveness of sitting time, typically >8 hours per day, provides many opportunities for intervention. Specific interventions are required to reduce sitting because it is such a habitual behavior and is reinforced by social norms and chair-dominant contexts.

In this pilot study, the investigators focus on three different types of prolonged sitting interruptions as variables. Studies have shown that frequent breaks in sitting may reduce risk for cardiometabolic disease. In older adults, the investigators anticipate that frequent sit-to-stand transitions will impact metabolic, inflammatory and other biomarkers, in particular those related to mitochondrial and endothelial function. A key limitation of previous sedentary intervention studies is that they have not impacted frequency of sit-to-stand transitions; rather, they decreased total sitting and increased standing time. Further, previous sedentary intervention studies have not directly compared frequent sit-to-stand transition interruptions with other interruption modalities associated with less frequent sit-to-stand transitions, for example, reduced overall sitting time (standing more) or with occasional walking breaks. The investigators propose to test these sedentary behavior interruptions modalities to disrupt prolonged sitting and explore mitochondrial- and endothelial function-based mechanisms of action. Biologic theories suggest that interrupting sitting via sit-to-stand muscle contraction and increased blood flow to extremities is key to improving in healthy aging outcomes.

In a controlled laboratory study of prolonged sitting, 3 different interruption break types will be utilized. Ten sedentary, postmenopausal participants 55+ years of age and body mass index (BMI) of 27-45 will be enrolled. After screening and enrollment, participants will visit the clinic on 4 occasions for a 6-hour monitoring period and, following a 1-hour sitting run-in period, complete each of 4 5-hour sitting protocols. The 3 sitting interruption protocols will each include sitting interruptions of different break frequency and type and will allow evaluation of the effect of sit-to-stand transitions and interruption type on acute metabolism and health outcomes. All study protocols include baseline, mid-point, and end-of-study bathroom breaks for urine sample collection with additional bathroom breaks allowed as needed. During each protocol at multiple time points, blood samples will be collected to assess changes in biomarkers of glycemic regulation (glucose and insulin areas under the curve) and mitochondrial function over the course of the sitting protocols. During each protocol at multiple time points, changes in endothelial function, specifically, blood pressure (indirect measure) and femoral flow-mediated dilation (direct measure), will be assessed. Changes in these measures will be compared between protocols. A small aliquot (0.5mL) of plasma samples and urine samples collected during the protocol will be banked for possible ancillary, exploratory studies. This study is a crossover design and each participant will be her own control. The investigators hypothesize that frequent sit-to-stands during a 5-hour sitting period will result in health benefits that can be observed with a simple 2-minute standing interruption, and that this will be associated with improvements in metabolism and endothelial function. The investigators will test this hypothesis in the following aim:

Study Aim: Using a randomized, controlled crossover study design, assess the feasibility and metabolic and endothelial function outcomes of an acute bout of prolonged sitting ± standing or walking interruptions using targeted metabolic and endothelial function biomarker analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal woman, any ethnicity/race, 55+ years of age.
2. Ambulatory, medically stable, able to give informed consent, and safely complete the protocols.
3. Fluent in the English language.
4. Body Mass Index range of 27-45kg/m2.
5. Sedentary: Average ≥6hr sitting time, and <20min physical activity on 3 or more days per week, as assessed by self report.

Exclusion Criteria:

1. Mental states that would preclude complete understanding of the protocol and compliance.
2. Chronic illness that may be associated with weight change (HIV/AIDS, active cancer, or uncontrolled thyroid disease).
3. Body Mass Index <27 or >45kg/m2.
4. Anemia (hemoglobin ≤11g/dL) - determined by CBC test done at screening.
5. Arthritis or degenerative joint disease affecting knees where repeated sitting/standing interruptions might cause pain.
6. Personal or family history of venous thrombosis.
7. Type 1 diabetes mellitus
8. Poorly controlled hypertension (SBP ≥165 or DBP ≥100).
9. Weight instability in past 3 months (no more than 5% up or down).
10. Participants <65 years of age with HbA1c ≥53 mmol/mol (7%) and participants ≥65 years of age with HbA1c ≥58mmol/mol (7.5%) will be excluded for uncontrolled diabetes.34,35
11. Use of insulin medications.
12. Regular use of vasodilator medication AND high risk of stroke and/or heart attack (i.e., history of multiple hospitalizations (>2X in the last 6 months), congestive heart failure, atrial fibrillation, and/or stroke).
13. Use of any immunosuppressant or corticosteroid medication.
14. Use of medications that might cause weight change (e.g., second generation anti-psychotics).
15. < 6hr average daily sitting time.

17) ≥20min physical activity average on 3 or more days per week 18) Participating in another clinical trial. 19) Blood donation less than 56 days prior to screening visit. 20) Smoking cigarettes or anything, and other use of tobacco products.

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in endothelial function | Five hours
  Change in endothelial function will be assessed by femoral flow-mediated dilation (FMD) and blood pressure measurements collected during the course of each study visit condition. Intervention-induced change will be compared to change observed during the control condition.
Change in glycemic regulation | Five hours
  Change in glycemic regulation will be assessed by measuring plasma glucose and insulin concentrations in blood collected at 30-min intervals during each study visit condition. Intervention-induced change will be compared to change observed during the control condition.

SECONDARY OUTCOMES:
Study feasibility | 3 months
  Feasibility will be assess by tabulating the following: number of recruitment inquiries, number of participants screened at clinic, number of participants enrolled, number of participants completing all protocols, and acceptability of sitting protocols to participants.
Change in mitochondrial metabolites | Five hours
  Change in mitochondrial metabolites will be assessed by mass spectrometry measurements of plasma samples collected at the beginning and end of each study visit condition. Intervention-induced change will be compared to change observed during the control condition.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kerr J, Crist K, Vital DG, Dillon L, Aden SA, Trivedi M, Castellanos LR, Godbole S, Li H, Allison MA, Khemlina GL, Takemoto ML, Schenk S, Sallis JF, Grace M, Dunstan DW, Natarajan L, LaCroix AZ, Sears DD. Acute glucoregulatory and vascular outcomes of three strategies for interrupting prolonged sitting time in postmenopausal women: A pilot, laboratory-based, randomized, controlled, 4-condition, 4-period crossover trial. PLoS One. 2017 Nov 30;12(11):e0188544. doi: 10.1371/journal.pone.0188544. eCollection 2017. PMID 29190761